CLINICAL TRIAL: NCT05331820
Title: Influence of Reminder on Enhancing Patient Compliance in Patients With Fixed Orthodontic Appliance Treatment (a Randomized Controlled Clinical Trial)
Brief Title: The Influence of Weekly Reminders on Enhancing Patient Compliance in Patients With Fixed Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shara Qadir Hussein (Other)
Responsible Party: Sponsor-Investigator, Shara Qadir Hussein, investigator, University of Sulaimani
Organization: University of Sulaimani (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2021-12-03; First posted 2022-04-18 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Patient Compliance
Keywords: patient compliance; orthodontic patients; reminder
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: the orthodontist did not know the group of their patients .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care group (No Intervention): this group of participants will be used to compare to the intervention group. normal and professional instructions and motivation will be given to them but they will not receive weekly reminders about the importance of adherence to instructions
- weekly reminder group (Experimental): this group of participants will receive a weekly reminder about the importance of oral hygiene, appliance care, and adherence to recommendations from the dentist.
  Interventions: Other: weekly mobile reminder

INTERVENTIONS:
Other: weekly mobile reminder — a weekly reminder will be sent to participants in the intervention group via mobile internet applications
  Arms: weekly reminder group

SUMMARY:
this study is a randomized clinical trial to evaluate the effect of sending weekly reminders to patients undergoing fixed orthodontic appliance treatment. two groups will be formed and participants of the study will be divided between the two groups randomly. the intervention group will receive weekly reminders about the importance of oral hygiene and appliance care with adherence to scheduled appointments. the difference between these parameters will be evaluated between the control and intervention groups to describe the importance of weekly reminders to enhance the compliance and cooperation of the patient. the oral hygiene of the patient will include plaque level(plaque index), gingival statue level( bleeding index), and white spot lesion . appliance care will be recorded when in case of bracket failure and appointments missed will also be recorded .

ELIGIBILITY:
Inclusion Criteria:

* Patients with a fixed orthodontic appliance
* both gender
* age 15-25 years old
* patient or parent have smartphone and internet connection
* malocclusion of the patient undergoing treatment according to Index of Orthodontic Treatment Need IOTN should be grade 1,2, and 3
* good gingival health.

Exclusion Criteria:

* Patients with a removable appliance
* cleft lip and palate patients
* patients with hypomineralization visible on anterior teeth
* susceptible to periodontal disease
* have diabetes
* handicap patients, a severe malocclusion above IOTN grade 3, ceramic brackets, and a child with parents that cannot read.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2021-11-28 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
oral hygiene examination The plaque index system | during the intervention ( follow up for 6 months )
  consists of 4 degree higher score is the worst situation and 0 is the best
oral hygiene examination - Bleeding Index | during the intervention ( follow up for 6 months )
  bleeding on probing . conatains 3 scores 0 - no bleeding
  1. bleeding after 30 seconds
  2. bleeding immediately score 0 is the best and score 2 is the worst
oral hygiene examination white spot lesion | during the intervention ( follow up for 6 months )
  white spot lesion on the tooth will be examined clinically and recorded in photographs
appliance care | during the intervention ( follow up for 6 months )
  bracket failure will be recorded if there is any brackets/"
  ] bracket fracture will be recorded at appointments if there is any bracket dislodgments that needs replacement
adherence to appointment | during the intervention ( follow up for 6 months
  if patient does not come to the appointment it will be recorded as lack of adherence to appointments .

CONTACTS AND LOCATIONS:
Overall Officials: Hadi M Ismail, as.professor, Principal Investigator — University of Sulaimani
Locations (1):
- University of Sulaimani, Sulaymaniyah, Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: No
The initial follow up period for this research is 6 months , if participants agree it may be increased to use in other research for longer follow up.

REFERENCES:
- [Background] Mohammed H, Rizk MZ, Wafaie K, Ulhaq A, Almuzian M. Reminders improve oral hygiene and adherence to appointments in orthodontic patients: a systematic review and meta-analysis. Eur J Orthod. 2019 Mar 29;41(2):204-213. doi: 10.1093/ejo/cjy045. PMID 29947755
- [Background] Lima IFP, de Andrade Vieira W, de Macedo Bernardino I, Costa PA, Lima APB, Pithon MM, Paranhos LR. Influence of reminder therapy for controlling bacterial plaque in patients undergoing orthodontic treatment: A systematic review and meta-analysis. Angle Orthod. 2018 Jul;88(4):483-493. doi: 10.2319/111117-770.1. Epub 2018 Apr 17. PMID 29664334
- [Derived] Hussein S, Ismail H. Influence of Reminder on Enhancing Compliance in Patients with Fixed Orthodontic Appliance Treatment (a Randomized Controlled Clinical Trial). Patient Prefer Adherence. 2023 Jul 20;17:1759-1769. doi: 10.2147/PPA.S418109. eCollection 2023. PMID 37492635